CLINICAL TRIAL: NCT03432832
Title: Emotion Awareness and Skills Enhancement (EASE) Program: A Clinical Trial
Brief Title: Emotion Awareness and Skills Enhancement Program
Acronym: EASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Carla Mazefsky, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20110317
Record Dates: First submitted 2018-01-17; First posted 2018-02-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: per protocol analysis versus intent to treat analytic approach due to the pandemic
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Awareness/Skills Enhancement (Experimental): EASE Therapy includes 16 weekly sessions focused on mindfulness exercise, review of prior content, practicing prior skills, outline of current session, discussion of the new skill, handouts, practice and plan for out of session practice held in Webster Hall in Pittsburgh, at the Center for the Prevention of Youth Behavior Problems in Tuscaloosa or via telehealth conferencing software. The investigators will apply a multimodal teaching approach, where individual therapy is buttressed by parent involvement and practice sessions in the youth's community. A secure website developed for this project (emotion-Coach or "e-Coach") will augment the intervention by providing online supports to increase treatment intensity or dosage. There will be specific information on how to reinforce the skills at home and in the community.
  Interventions: Behavioral: EASE
- Supportive Therapy (Active Comparator): Supportive Therapy will involve attending 16 weekly therapy sessions held in Webster Hall in Pittsburgh, at the Center for the Prevention of Youth Behavior Problems in Tuscaloosa or via telehealth conferencing software. The intervention will not involve mindfulness or other emotion regulation strategies used in EASE. The therapy will be tailored to the individual's needs and will include aspects common in supportive therapy such as reflective listening, antecedent management, and problem-solving. This program does not have an online component.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: EASE — Weekly behavioral sessions with therapist to work on emotional control through measures such as mindfulness.
  Arms: Emotion Awareness/Skills Enhancement
Behavioral: Supportive Therapy — Weekly behavioral sessions with a therapist to work on emotional control
  Arms: Supportive Therapy

SUMMARY:
This project will address impaired emotion regulation in adolescents with ASD (autism spectrum disorder). There are no evidence-based interventions to improve emotion regulation (ER) in this population, yet poor emotion regulation often leads to maladaptive behavior and substantially impedes capacity to learn and function across all life settings, and reduce their quality of life and that of their families. The primary objective of this study is to formally evaluate efficacy of EASE via a sufficiently powered, two-site randomized-controlled trial (RCT).

DETAILED DESCRIPTION:
The current study is to test a new intervention called Emotional Awareness and Skills Enhancement (EASE). This program was designed to address ASD-specific obstacles to effective emotion regulation, such as reduced awareness concerning others' intentions, a limited repertoire of behavioral responses, and inadequate language for understanding emotional experiences. This new program is based on an acceptance-based approach in which awareness of emotion is developed, emotions (whether negative or positive) are accepted, and behavior is regulated in the face of intense emotion. The goal is not to learn to avoid negative emotions, but rather to develop a collection of abilities which allow the individual to manage stress and act in ways that are more adaptive. The investigators expect to find that participants' emotion dysregulation will decrease and their adaptive function will increase following completion of the EASE program.

ELIGIBILITY:
Inclusion Criteria:

1. ages 12-21 years, inclusive
2. A diagnosis of ASD (autism spectrum disorder), as defined by exceeding the ASD cutoff on the ADOS-2 (Autism Diagnostic Observation Scale) or ADI-R (Autism Diagnostic Interview-Revised) In. If the participant has completed the ADOS in a previous study within 3 years and signs a release of information to obtain it, they will not be required to complete another ADOS.
3. Average verbal intellectual ability (Wechsler Abbreviated Scale of Intelligence-2 [WASI-2] FSIQ >=75).
4. Fluent in the English language
5. Problems with regulating emotions based on parent report 6) Parent/guardian who will attend sessions and assessments.

Exclusion Criteria:

1. Current concerns of suicidality that warrants immediate clinical care (such potential participants will be referred elsewhere for treatment), determined by clinical interview.
2. Previous or current diagnosis of a psychotic disorder.
3. Receiving concurrent psychotherapy treatment for emotional issues (i.e., depression, anxiety, anger) that overlaps with the current study. This will be assessed using current treatment items on the demographic forms.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The Clinical Global Impression Scale- Improvement (CGI-I) | The CGI-I will be completed at 16 weeks (post-treatment)
  The CGI-I will be used as a measure of overall improvement. The CGI-I (Improvement) scale was designed to measure overall symptomatic change at a specific time as compared to baseline that is completed by a rater who is blind to treatment assignment. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse). It is only a single item, and lower scores indicate more improvement.
Emotion Dysregulation Inventory Reactivity Scale Short Form (EDI-SF) | The EDI-SF will be completed at 16 weeks (post-treatment).
  The EDI SF is a measure of emotional reactivity and regulation. The EDI SF is based on theta scores, with a mean of 0 and SD of 1 and possible range from -1.99 to 2.105. Higher scores suggest greater dysregulation, so improvement would be measured by a decrease in scores.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | The CGI-I will be completed at 16 weeks (post-treatment)
  The Brief Psychiatric Rating Scale (BPRS) is an interview-based measure of psychopathology severity widely used in clinical trials. It consists of 24 items that measure psychiatric symptoms, each of which are on a 1 (not reported) to 7 (very severe) scale, so that lower scores are an indication of improvement. An assignment naïve rater scores the items based upon client report and clinical observation. All scales ask about symptoms over the last 7 days. The single item on "Global Improvement" will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Mazefsky, PhD, Principal Investigator — University of Pittsburgh; Susan White, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama, Tuscaloosa, Alabama
  - Shannondora Porton, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abidin, R. R. (2012). Parenting Stress Index, Fourth Edition Short Form (PSI-4). Lutz, FL: PAR.
- [Background] Achenbach, T. M., & Rescorla, L. (2001). Manual for the ASEBA school-age forms and profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Aldao A, Nolen-Hoeksema S, Schweizer S. Emotion-regulation strategies across psychopathology: A meta-analytic review. Clin Psychol Rev. 2010 Mar;30(2):217-37. doi: 10.1016/j.cpr.2009.11.004. Epub 2009 Nov 20. PMID 20015584
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Aman M, Rettiganti M, Nagaraja HN, Hollway JA, McCracken J, McDougle CJ, Tierney E, Scahill L, Arnold LE, Hellings J, Posey DJ, Swiezy NB, Ghuman J, Grados M, Shah B, Vitiello B. Tolerability, Safety, and Benefits of Risperidone in Children and Adolescents with Autism: 21-Month Follow-up After 8-Week Placebo-Controlled Trial. J Child Adolesc Psychopharmacol. 2015 Aug;25(6):482-93. doi: 10.1089/cap.2015.0005. PMID 26262903
- [Background] Anagnostou E, Jones N, Huerta M, Halladay AK, Wang P, Scahill L, Horrigan JP, Kasari C, Lord C, Choi D, Sullivan K, Dawson G. Measuring social communication behaviors as a treatment endpoint in individuals with autism spectrum disorder. Autism. 2015 Jul;19(5):622-36. doi: 10.1177/1362361314542955. Epub 2014 Aug 5. PMID 25096930
- [Background] Anderson DK, Liang JW, Lord C. Predicting young adult outcome among more and less cognitively able individuals with autism spectrum disorders. J Child Psychol Psychiatry. 2014 May;55(5):485-94. doi: 10.1111/jcpp.12178. Epub 2013 Dec 9. PMID 24313878
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Baker AE, Lane A, Angley MT, Young RL. The relationship between sensory processing patterns and behavioural responsiveness in autistic disorder: a pilot study. J Autism Dev Disord. 2008 May;38(5):867-75. doi: 10.1007/s10803-007-0459-0. PMID 17899349
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Baskin TW, Tierney SC, Minami T, Wampold BE. Establishing specificity in psychotherapy: a meta-analysis of structural equivalence of placebo controls. J Consult Clin Psychol. 2003 Dec;71(6):973-9. doi: 10.1037/0022-006X.71.6.973. PMID 14622072
- [Background] Bishop-Fitzpatrick L, Minshew NJ, Eack SM. A systematic review of psychosocial interventions for adults with autism spectrum disorders. J Autism Dev Disord. 2013 Mar;43(3):687-94. doi: 10.1007/s10803-012-1615-8. PMID 22825929
- [Background] Boulter C, Freeston M, South M, Rodgers J. Intolerance of uncertainty as a framework for understanding anxiety in children and adolescents with autism spectrum disorders. J Autism Dev Disord. 2014 Jun;44(6):1391-402. doi: 10.1007/s10803-013-2001-x. PMID 24272526
- [Background] Carroll D, Hallett V, McDougle CJ, Aman MG, McCracken JT, Tierney E, Arnold LE, Sukhodolsky DG, Lecavalier L, Handen BL, Swiezy N, Johnson C, Bearss K, Vitiello B, Scahill L. Examination of aggression and self-injury in children with autism spectrum disorders and serious behavioral problems. Child Adolesc Psychiatr Clin N Am. 2014 Jan;23(1):57-72. doi: 10.1016/j.chc.2013.08.002. PMID 24231167
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193
- [Background] Chiesa A, Serretti A, Jakobsen JC. Mindfulness: top-down or bottom-up emotion regulation strategy? Clin Psychol Rev. 2013 Feb;33(1):82-96. doi: 10.1016/j.cpr.2012.10.006. Epub 2012 Oct 23. PMID 23142788
- [Background] Connor-Smith JK, Compas BE, Wadsworth ME, Thomsen AH, Saltzman H. Responses to stress in adolescence: measurement of coping and involuntary stress responses. J Consult Clin Psychol. 2000 Dec;68(6):976-92. PMID 11142550
- [Background] Constantino JN, Abbacchi AM, Lavesser PD, Reed H, Givens L, Chiang L, Gray T, Gross M, Zhang Y, Todd RD. Developmental course of autistic social impairment in males. Dev Psychopathol. 2009 Winter;21(1):127-38. doi: 10.1017/S095457940900008X. PMID 19144226
- [Background] Croen LA, Najjar DV, Ray GT, Lotspeich L, Bernal P. A comparison of health care utilization and costs of children with and without autism spectrum disorders in a large group-model health plan. Pediatrics. 2006 Oct;118(4):e1203-11. doi: 10.1542/peds.2006-0127. PMID 17015508
- [Background] Croen LA, Zerbo O, Qian Y, Massolo ML, Rich S, Sidney S, Kripke C. The health status of adults on the autism spectrum. Autism. 2015 Oct;19(7):814-23. doi: 10.1177/1362361315577517. Epub 2015 Apr 24. PMID 25911091
- [Background] Crone EA, Dahl RE. Understanding adolescence as a period of social-affective engagement and goal flexibility. Nat Rev Neurosci. 2012 Sep;13(9):636-50. doi: 10.1038/nrn3313. PMID 22903221
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Denissen JJ, Penke L, Schmitt DP, van Aken MA. Self-esteem reactions to social interactions: evidence for sociometer mechanisms across days, people, and nations. J Pers Soc Psychol. 2008 Jul;95(1):181-96. doi: 10.1037/0022-3514.95.1.181. PMID 18605859
- [Background] Eack SM, Greenwald DP, Hogarty SS, Bahorik AL, Litschge MY, Mazefsky CA, Minshew NJ. Cognitive enhancement therapy for adults with autism spectrum disorder: results of an 18-month feasibility study. J Autism Dev Disord. 2013 Dec;43(12):2866-77. doi: 10.1007/s10803-013-1834-7. PMID 23619953
- [Background] Eaves LC, Ho HH. Young adult outcome of autism spectrum disorders. J Autism Dev Disord. 2008 Apr;38(4):739-47. doi: 10.1007/s10803-007-0441-x. Epub 2007 Sep 1. PMID 17764027
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474
- [Background] Gerdts J, Bernier R. The broader autism phenotype and its implications on the etiology and treatment of autism spectrum disorders. Autism Res Treat. 2011;2011:545901. doi: 10.1155/2011/545901. Epub 2011 Aug 17. PMID 22937250
- [Background] Gotham K, Brunwasser SM, Lord C. Depressive and anxiety symptom trajectories from school age through young adulthood in samples with autism spectrum disorder and developmental delay. J Am Acad Child Adolesc Psychiatry. 2015 May;54(5):369-76.e3. doi: 10.1016/j.jaac.2015.02.005. Epub 2015 Feb 17. PMID 25901773
- [Background] Gotink RA, Chu P, Busschbach JJ, Benson H, Fricchione GL, Hunink MG. Standardised mindfulness-based interventions in healthcare: an overview of systematic reviews and meta-analyses of RCTs. PLoS One. 2015 Apr 16;10(4):e0124344. doi: 10.1371/journal.pone.0124344. eCollection 2015. PMID 25881019 (Retraction: PMID 30978236 PLoS One. 2019 Apr 12;14(4):e0215608)
- [Background] Greco LA, Baer RA, Smith GT. Assessing mindfulness in children and adolescents: development and validation of the Child and Adolescent Mindfulness Measure (CAMM). Psychol Assess. 2011 Sep;23(3):606-14. doi: 10.1037/a0022819. PMID 21480722
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Guy L, Souders M, Bradstreet L, DeLussey C, Herrington JD. Brief report: emotion regulation and respiratory sinus arrhythmia in autism spectrum disorder. J Autism Dev Disord. 2014 Oct;44(10):2614-20. doi: 10.1007/s10803-014-2124-8. PMID 24752681
- [Background] Hodges K, Kim CS. Psychometric study of the Child and Adolescent Functional Assessment Scale: prediction of contact with the law and poor school attendance. J Abnorm Child Psychol. 2000 Jun;28(3):287-97. doi: 10.1023/a:1005100521818. PMID 10885686
- [Background] Howlin P, Goode S, Hutton J, Rutter M. Adult outcome for children with autism. J Child Psychol Psychiatry. 2004 Feb;45(2):212-29. doi: 10.1111/j.1469-7610.2004.00215.x. PMID 14982237
- [Background] Ives-Deliperi VL, Solms M, Meintjes EM. The neural substrates of mindfulness: an fMRI investigation. Soc Neurosci. 2011;6(3):231-42. doi: 10.1080/17470919.2010.513495. Epub 2010 Sep 9. PMID 20835972
- [Background] Khor AS, Melvin GA, Reid SC, Gray KM. Coping, daily hassles and behavior and emotional problems in adolescents with high-functioning autism/Asperger's Disorder. J Autism Dev Disord. 2014 Mar;44(3):593-608. doi: 10.1007/s10803-013-1912-x. PMID 23933998
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Mazefsky CA, Minshew NJ. The spectrum of autism-from neuronal connections to behavioral expression. Virtual Mentor. 2010 Nov 1;12(11):867-72. doi: 10.1001/virtualmentor.2010.12.11.cprl1-1011. PMID 23186793
- [Background] Mazefsky CA, Conner CM, Oswald DP. Association between depression and anxiety in high-functioning children with autism spectrum disorders and maternal mood symptoms. Autism Res. 2010 Jun;3(3):120-7. doi: 10.1002/aur.133. PMID 20578069
- [Background] Mazefsky CA, Borue X, Day TN, Minshew NJ. Emotion regulation patterns in adolescents with high-functioning autism spectrum disorder: comparison to typically developing adolescents and association with psychiatric symptoms. Autism Res. 2014 Jun;7(3):344-54. doi: 10.1002/aur.1366. Epub 2014 Mar 7. PMID 24610869
- [Background] Mazefsky CA, Day TN, Siegel M, White SW, Yu L, Pilkonis PA; Autism and Developmental Disabilities Inpatient Research Collaborative (ADDIRC). Development of the Emotion Dysregulation Inventory: A PROMIS(R)ing Method for Creating Sensitive and Unbiased Questionnaires for Autism Spectrum Disorder. J Autism Dev Disord. 2018 Nov;48(11):3736-3746. doi: 10.1007/s10803-016-2907-1. PMID 27699685
- [Background] Mazefsky CA, White SW. Emotion regulation: concepts & practice in autism spectrum disorder. Child Adolesc Psychiatr Clin N Am. 2014 Jan;23(1):15-24. doi: 10.1016/j.chc.2013.07.002. Epub 2013 Aug 30. PMID 24231164
- [Background] McCracken JT, McGough J, Shah B, Cronin P, Hong D, Aman MG, Arnold LE, Lindsay R, Nash P, Hollway J, McDougle CJ, Posey D, Swiezy N, Kohn A, Scahill L, Martin A, Koenig K, Volkmar F, Carroll D, Lancor A, Tierney E, Ghuman J, Gonzalez NM, Grados M, Vitiello B, Ritz L, Davies M, Robinson J, McMahon D; Research Units on Pediatric Psychopharmacology Autism Network. Risperidone in children with autism and serious behavioral problems. N Engl J Med. 2002 Aug 1;347(5):314-21. doi: 10.1056/NEJMoa013171. PMID 12151468
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] Rieffe C, De Bruine M, De Rooij M, Stockmann L. Approach and avoidant emotion regulation prevent depressive symptoms in children with an Autism Spectrum Disorder. Int J Dev Neurosci. 2014 Dec;39:37-43. doi: 10.1016/j.ijdevneu.2014.06.003. Epub 2014 Jun 19. PMID 24951836
- [Background] Shallcross AJ, Gross JJ, Visvanathan PD, Kumar N, Palfrey A, Ford BQ, Dimidjian S, Shirk S, Holm-Denoma J, Goode KM, Cox E, Chaplin W, Mauss IB. Relapse prevention in major depressive disorder: Mindfulness-based cognitive therapy versus an active control condition. J Consult Clin Psychol. 2015 Oct;83(5):964-75. doi: 10.1037/ccp0000050. Epub 2015 Aug 10. PMID 26371618
- [Background] Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: prevalence, comorbidity, and associated factors in a population-derived sample. J Am Acad Child Adolesc Psychiatry. 2008 Aug;47(8):921-9. doi: 10.1097/CHI.0b013e318179964f. PMID 18645422
- [Background] Taylor JL, Mailick MR. A longitudinal examination of 10-year change in vocational and educational activities for adults with autism spectrum disorders. Dev Psychol. 2014 Mar;50(3):699-708. doi: 10.1037/a0034297. Epub 2013 Sep 2. PMID 24001150
- [Background] Verheij C, Louwerse A, van der Ende J, Eussen ML, Van Gool AR, Verheij F, Verhulst FC, Greaves-Lord K. The Stability of Comorbid Psychiatric Disorders: A 7 Year Follow Up of Children with Pervasive Developmental Disorder-Not Otherwise Specified. J Autism Dev Disord. 2015 Dec;45(12):3939-48. doi: 10.1007/s10803-015-2592-5. PMID 26456972
- [Background] White SW, Albano AM, Johnson CR, Kasari C, Ollendick T, Klin A, Oswald D, Scahill L. Development of a cognitive-behavioral intervention program to treat anxiety and social deficits in teens with high-functioning autism. Clin Child Fam Psychol Rev. 2010 Mar;13(1):77-90. doi: 10.1007/s10567-009-0062-3. PMID 20091348
- [Background] White SW, Ollendick T, Albano AM, Oswald D, Johnson C, Southam-Gerow MA, Kim I, Scahill L. Randomized controlled trial: Multimodal Anxiety and Social Skill Intervention for adolescents with autism spectrum disorder. J Autism Dev Disord. 2013 Feb;43(2):382-94. doi: 10.1007/s10803-012-1577-x. PMID 22735897
- [Background] White SW, Elias R, Salinas CE, Capriola N, Conner CM, Asselin SB, Miyazaki Y, Mazefsky CA, Howlin P, Getzel EE. Students with autism spectrum disorder in college: Results from a preliminary mixed methods needs analysis. Res Dev Disabil. 2016 Sep;56:29-40. doi: 10.1016/j.ridd.2016.05.010. Epub 2016 Jun 1. PMID 27262124
- [Background] White SW, Elias R, Capriola-Hall NN, Smith IC, Conner CM, Asselin SB, Howlin P, Getzel EE, Mazefsky CA. Development of a College Transition and Support Program for Students with Autism Spectrum Disorder. J Autism Dev Disord. 2017 Oct;47(10):3072-3078. doi: 10.1007/s10803-017-3236-8. PMID 28685409
- [Derived] White SW, Conner CM, Beck K, Mazefsky CA. Efficacy of the Emotion Awareness and Skills Enhancement (EASE) Program in Autism: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2025 Jul 31:S0890-8567(25)01410-8. doi: 10.1016/j.jaac.2025.07.1058. Online ahead of print. PMID 40750084

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03432832/Prot_SAP_000.pdf